CLINICAL TRIAL: NCT07342686
Title: A Hypothalamic Injury-Stratified Nursing Care Pathway for Pediatric Craniopharyngioma Survivors: Advancing Nursing Leadership in Complex Chronic Disease Management
Brief Title: Hypothalamic-Stratified Nursing Pathway for Pediatric Craniopharyngioma
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Other Study IDs: WestChinaH-HX-2025-07
Record Dates: First submitted 2025-12-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2013-01

CONDITIONS: Craniopharyngioma; Growth Hormone Deficiency (GHD)
Keywords: Hypothalamic Injury; Neuropsychological Development; Stratified Nursing Pathway; Multicenter Retrospective Study
MeSH Terms: conditions — Craniopharyngioma; Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Grade 0: Hypothalamic Injury Uninvolved (n=100)
- Grade 1: Mild Compression (n=250)
- Grade 2: Significant Invasion (n=150)

SUMMARY:
The goal of this multicenter retrospective cohort study is to determine whether MRI-graded hypothalamic injury severity predicts growth-hormone deficiency (GHD) and neuropsychological morbidity in 500 children and adolescents (≤ 18 y) who underwent craniopharyngioma resection at six Chinese pediatric centers between 2013 and 2023 and were followed ≥ 2 years. The main questions it aims to answer are:

1. Does increasing hypothalamic injury grade (Grade 0 = uninvolved, Grade 1 = mild compression, Grade 2 = significant invasion) independently correlate with higher incidence of GHD, lower IGF-1 levels, greater height SDS decline, and increased need for recombinant human GH therapy?
2. Is higher injury grade associated with worse neuropsychological outcomes-lower IQ, impaired executive function, emotional disorders, and obesity-after adjustment for age, tumor size, and extent of resection?

Researchers compared the three injury-grade groups to quantify endocrine and neuro-behavioral outcomes and to catalog differentiated nursing needs (growth monitoring frequency, dietary-behavioral plans, psychological support intensity, comorbidity surveillance). Participants underwent pre- and post-operative MRI grading by blinded neuroradiologists, standardized endocrine stimulation tests, annual neuropsychological testing (WISC-IV, BRIEF, CBCL), and detailed nursing-documentation review; all data were analyzed with Spearman correlation, ANOVA, and multivariable logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤18 years at the time of craniopharyngioma resection;
* Pathologically confirmed craniopharyngioma;
* Postoperative follow-up duration ≥2 years;
* Complete preoperative and postoperative MRI data, endocrine test results, neuropsychological assessment records, and nursing documentation;
* No preoperative GHD, neuropsychological disorders, or other systemic diseases affecting growth or neurodevelopment.

Exclusion Criteria:

* Preoperative diagnosis of GHD, cognitive impairment, or emotional disorders;
* Concurrent intracranial tumors or systemic diseases (e.g., congenital growth hormone deficiency, Down syndrome);
* Loss to follow-up or incomplete clinical data;
* Tumor recurrence requiring reoperation during follow-up.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: **Study Population Description** Children and adolescents ≤ 18 years of age who underwent primary surgical resection for craniopharyngioma at one of six tertiary pediatric centers in China between January 2013 and December 2023, had complete pre- and post-operative brain MRI, endocrine, and neuropsychological data, and were followed for ≥ 2 years without tumor re-operation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of growth hormone deficiency (GHD) at 2 years post-surgery | 2 years
  defined as peak GH < 10 ng/mL on stimulation testing plus age-/sex-adjusted IGF-1 below reference range

SECONDARY OUTCOMES:
Change in height standard-deviation score (Δ-height SDS) from baseline to final follow-up. | 2 years
Proportion of patients who initiate recombinant human GH (rhGH) therapy | 2 years
Normalized IGF-1 level (age-/sex-adjusted z-score) at final follow-up. | 2 years
Mean full-scale IQ score (WISC-IV) and rate of cognitive impairment (IQ < 85). | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol